CLINICAL TRIAL: NCT02754791
Title: Reducing Blood Culture Contamination: a Prospective Crossover Study
Brief Title: Reducing Blood Culture Contamination:
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Shaare Zedek Medical Center (Other)
Collaborators: Magnolia Medical Technologies, Inc. (Industry); 3M (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None
Other Study IDs: 42/16
Record Dates: First submitted 2016-04-19; First posted 2016-04-28 (Estimated); Last update posted 2016-05-03 (Estimated); Status verified 2016-05

CONDITIONS: Preventing Blood Culture Contamination

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- Monthly report (No Intervention): A monthly report will be submitted to department heads describing their departments rate of blood culture contamination and comparing it to blood culture contamination rate in previous months and to blood culture contamination rate of the hospital as a whole
- Steripath (Experimental): The Steripath device (Magnolia) will be used to take blood cultures in this arm instead of standard methods. This will be in addition to a departmental monthly report (described above).
  Interventions: Device: Steripath
- Soluprep wipes (Experimental): In this arm, skin sterilization will be achieved using Soluprep wipes (3M) instead of standard methods (alcohol wipes).This will be in addition to a departmental monthly report (described above).
  Interventions: Device: Soluprep

INTERVENTIONS:
Device: Steripath — A device that diverts the first 2 ml of blood drawn in order to reduce contamination
  Arms: Steripath
Device: Soluprep — Wipes containing alcohol (70%) and chlorhexidine (2%) to achieve skin sterilization
  Arms: Soluprep wipes

SUMMARY:
Bloodstream infections cause significant morbidity and mortality and their prompt identification is an essential part of modern medicine. False positive results in blood cultures are primarily due to contaminants. It has been estimated that up to 50% of positive blood cultures represent contamination. These false positive cultures, at the microbiological laboratory level, require significant additional resources for workup. Additionally, they result in unnecessary antibiotic treatment and hospitalization days, causing needless harm to patients. Various methods have been implemented in order to reduce blood culture contaminants, including modifying the solution used for sterilizing the skin and feedback on contamination rates. However, it has been shown that the bacteria which colonize the human skin are not only on the surface but in fact colonize deeper surfaces as well. The SteriPath device diverts the initial 1-2 ml blood so as to remove any potential skin plug with contaminants. Thus, the principle object of this study is the determination of the rate of contamination of blood culture taken prior to initiating intervention versus the rate of contamination using three interventions: Monthly feedback via departmental report card, a chlorhexidine plus alcohol wipe and the SteriPath device. Secondary objectives will include ease of use of the wipes and the SteriPath device and an estimate of the sensitivity of SteriPath device use to true bacteremia. If the various interventions will be shown to reduce contamination, researchers will also attempt to estimate the financial effects of those reductions, comparing intervention cost to estimated savings related to reduced contamination.

ELIGIBILITY:
Inclusion Criteria:

* adult patients hospitalized in our institution in whom blood cultures are taken

Exclusion Criteria:

* none

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1500 (Estimated)
Dates: Start 2016-05; Primary Completion 2017-05 (Estimated); Study Completion 2017-05 (Estimated)

PRIMARY OUTCOMES:
Percentage of contaminated blood cultures relative to overall blood cultures as compared to percentage in historical and parallel control groups | 6 months

SECONDARY OUTCOMES:
Ease of use of SteriPath device as evaluated by resident physicians and phlebotomists using a questionaire | 6 months
Cost effectiveness of Steripath device and chlorhexidine wipes in measured as cost of devices in dollars versus reduction of cost in dollars associated with reduced blood culture contamination | 6 months

IPD SHARING:
Plan to Share IPD: Undecided